CLINICAL TRIAL: NCT01408407
Title: A Phase II Study Designed to Evaluate the Value of Alkagin Paste in the Prevention of Radiation Dermatitis for Patients Undergoing External Radiation Therapy
Brief Title: Alkagin Paste in the Prevention of Radiation Dermatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Te Vuong (Other)
Collaborators: Avario Healthcare Inc. (Industry)
Responsible Party: Sponsor-Investigator, Dr. Te Vuong, MD-Director Radiation Oncology, Sir Mortimer B. Davis - Jewish General Hospital
Organization: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11-052
Record Dates: First submitted 2011-08-02; First posted 2011-08-03 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Anus Neoplasms; Rectal Neoplasms; Urogenital Neoplasms
Keywords: Patients with anal canal, low rectal or gynecological cancer
MeSH Terms: conditions — Anus Neoplasms; Rectal Neoplasms; Urogenital Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: standard of care (Active Comparator): Patients will be asked to apply Aveeno cream twice a day starting the day of their treatment until two weeks after the end of their treatment
  Interventions: Other: Aveeno cream
- Arm B: standard of care plus Alkagin paste (Experimental): Patients will apply Alkagin Paste to the treatment area everyday one week before starting radiotherapy, throughout treatment and for two weeks post treatment. They will also perform standard of care skin treatment.
  Interventions: Other: Aveeno cream; Other: Alkagin paste

INTERVENTIONS:
Other: Aveeno cream — Apply cream on irradiated area twice a day
Other: Alkagin paste — Apply Alkagin paste three times a day.
  Arms: Arm B: standard of care plus Alkagin paste

SUMMARY:
The purpose of this study is to determine whether Alkagin paste is effective at preventing radiodermatitis in patients receiving external beam radiation therapy to the perineal area.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving a dose of 45 Gy or more with concomitant chemotherapy to the perineal skin (for treatment of anal canal, low rectal or gynecological cancer).
* Patients able to understand and sign an informed consent form.
* Patients that do not have active connective tissue disorders.
* Patients 18 years or older.
* Patients that did not receive any previous radiation.
* Patients that do not have any known allergy to any ingredients of the Alkagin Paste
* Patients need to be able to apply the creams themselves or have help with applying the creams.
* Patients who have been offered to purchase silver clear underpants but have refused

Exclusion Criteria:

* Patients that have a type V or type VI skin type according to the Fitzpatrick scale (because these patients will likely have less radiodermatitis and if they do, it will be harder to evaluate it)

The Fitzpatrick Scale:

* Type I (scores 0-7) White; very fair; freckles. Always burns, never tans
* Type II (scores 8-16) White; fair. Usually burns, tans with difficulty
* Type III (scores 17-25) Beige; very common. Sometimes mild burn, gradually tans
* Type IV (scores 25-30) Beige with a brown tint; typical Mediterranean Caucasian skin. Rarely burns, tans with ease
* Type V (scores over 30) Dark brown. Very rarely burns, tans very easily
* Type VI Black. Never burns, tans very easily

  2) Patients with an allergic reaction to Alkagin Paste

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-12; Primary Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Maximum skin toxicity | 7 weeks post beginning of radiation treatments
  The objective of this study is to determine the occurrence and degree of acute skin toxicity in patients receiving radical radiation therapy with preventive application of Alkagin Paste compared to patients treated with institutional standard skin care.

CONTACTS AND LOCATIONS:
Overall Officials: Te Vuong, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada